CLINICAL TRIAL: NCT00696007
Title: Neoadjuvant Chemotherapy Plus Nephroureterectomy for Locally Advanced Upper Tract Transitional Cell Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was unable to recruit subjects meeting the study requirements.
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-039
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Transitional Cell Carcinoma
Keywords: Upper GU Tract Transitional Cell Carinoma; Nephroureterectomy; Chemotherapy; Gemcitabine; Cisplatin
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Gemcitabine; Cisplatin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): A neoadjuvant chemotherapy (gemcitabine and cisplatin) regimen administered before surgery-nephroureterectomy for upper tract TCC
  Interventions: Drug: Gemcitabine and cisplatin
- 2 (Other): A retrospective cohort group (approximately 60 subjects) identified from an institutional cancer registry who have undergone a nephroureterectomy alone over the past five years
  Interventions: Other: Retrospective comparison

INTERVENTIONS:
Drug: Gemcitabine and cisplatin — Neoadjuvant chemotherapy (gemcitabine and cisplatin) administered before Nephroureterectomy.
  Chemotherapy regimen of three cycles of gemcitabine and cisplatin, dosed over a 3 month period Each cycle would consist of gemcitabine and cisplatin on day 1, with two other doses of gemcitabine on day 8 and day 15.
  Gemcitabine dosing would be 1,000 mg/m² and cisplatin would be dosed at 70 mg/m²
  Other Names: Neoadjuvant Chemotherapy
  Arms: 1
Other: Retrospective comparison — 60 retrospective historical cohort group of subjects who have undergone a radical nephroureterectomy over the past five years
  Arms: 2

SUMMARY:
The purpose of this study is to test the effectiveness, safety and side effects of two chemotherapy drugs (gemcitabine and cisplatin) when combined with surgery after chemotherapy for patients with upper urinary tract cancer. The hypothesis is that undergoing chemotherapy prior to surgery will have a beneficial effect on prognosis and may improve overall survival as in patients with bladder cancer, and will allow better tolerance of chemotherapy than if it were given after surgery.

DETAILED DESCRIPTION:
This study will look at improving overall survival of those undergoing nephroureterectomy for upper tract TCC (transitional cell carcinoma, comparing the pathological response of tumors treated with Neoadjuvant Chemotherapy (gemcitabine and cisplatin) before surgery. There have been reported studies of neoadjuvant chemotherapy in the treatment of upper tract TCC, there have been no studies to date that include the chemotherapy agents gemcitabine and cisplatin that are currently indicated in treating TCC of the bladder in the neoadjuvant and adjuvant setting. These agents have been proven to have a better overall safety profile and tolerability allowing more patients to complete their regimens. Secondarily, study will compare disease free overall survival among patients treated with neoadjuvant chemotherapy and surgery versus surgery alone. This study may elucidate the potential benefit of these agents when treating TCC of the upper tracts and may provide a survival advantage in this specific patient population as compared to a historical cohort.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-2
* Estimated GFR>60
* High grade TCC on initial biopsy
* Clinical stage T1-T3, Nx, Mx based on the AJCC Classification system
* TCC confined to the ureter or renal pelvis
* Grade II neuropathy or less

Exclusion Criteria:

* Any other malignancy over the previous five years with a risk of relapse that exceeds 30%
* History of previous cystectomy
* Evidence of metastatic disease
* History of pelvic irradiation or prior chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Neoadjuvant chemotherapy (Gemcitabine and Cisplatin) Regime (3 cycles) before Nephroureterectomy | 5 years: follow ups 1st year/every 4 mths, 2nd & 3rd year to every 6 months, 4th & 5th yr-annually for patients who remain disease free

SECONDARY OUTCOMES:
Overall survival compared to institutional historical cohort of subjects who have undergone a nephroureterectomy alone. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G. Tretter, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Splinter TA, Pavone-Macaluso M, Jacqmin D, Roberts JT, Carpentier P, de Pauw M, Sylvester R. A European Organization for Research and Treatment of Cancer--Genitourinary Group phase 2 study of chemotherapy in stage T3-4N0-XM0 transitional cell cancer of the bladder: evaluation of clinical response. J Urol. 1992 Dec;148(6):1793-6. doi: 10.1016/s0022-5347(17)37031-3. PMID 1433610
- [Background] Raman JD, Sosa RE, Vaughan ED Jr, Scherr DS. Pathologic features of bladder tumors after nephroureterectomy or segmental ureterectomy for upper urinary tract transitional cell carcinoma. Urology. 2007 Feb;69(2):251-4. doi: 10.1016/j.urology.2006.09.065. PMID 17320658
- [Background] Brown GA, Busby JE, Wood CG, Pisters LL, Dinney CP, Swanson DA, Grossman HB, Pettaway CA, Munsell MF, Kamat AM, Matin SF. Nephroureterectomy for treating upper urinary tract transitional cell carcinoma: Time to change the treatment paradigm? BJU Int. 2006 Dec;98(6):1176-80. doi: 10.1111/j.1464-410X.2006.06524.x. PMID 17125474
- [Background] Keeley FX, Kulp DA, Bibbo M, McCue PA, Bagley DH. Diagnostic accuracy of ureteroscopic biopsy in upper tract transitional cell carcinoma. J Urol. 1997 Jan;157(1):33-7. PMID 8976209
- [Background] Hall MC, Womack S, Sagalowsky AI, Carmody T, Erickstad MD, Roehrborn CG. Prognostic factors, recurrence, and survival in transitional cell carcinoma of the upper urinary tract: a 30-year experience in 252 patients. Urology. 1998 Oct;52(4):594-601. doi: 10.1016/s0090-4295(98)00295-7. PMID 9763077
- [Background] Grossman HB, Natale RB, Tangen CM, Speights VO, Vogelzang NJ, Trump DL, deVere White RW, Sarosdy MF, Wood DP Jr, Raghavan D, Crawford ED. Neoadjuvant chemotherapy plus cystectomy compared with cystectomy alone for locally advanced bladder cancer. N Engl J Med. 2003 Aug 28;349(9):859-66. doi: 10.1056/NEJMoa022148. PMID 12944571
- [Background] Igawa M, Urakami S, Shiina H, Kishi H, Himeno Y, Ishibe T, Kadena H, Usui T. Neoadjuvant chemotherapy for locally advanced urothelial cancer of the upper urinary tract. Urol Int. 1995;55(2):74-7. doi: 10.1159/000282755. PMID 8533199